CLINICAL TRIAL: NCT06925685
Title: Long Term Follow up Study for Participants Treated With an Allogeneic CAR T-Cell Product in a Prior Clinical Study
Brief Title: Follow-Up for Study Participants Treated With an Allogeneic CAR T-Cell Product
Status: Enrolling by invitation | Type: Observational
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-LTFU-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Malignancies; Solid Tumors
Keywords: CAR T; Allogeneic CAR T; long term follow up
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational, long-term follow up (LTFU) study of participants who received an allogeneic CAR T product in a prior clinical study. Participants will be followed for 15 years after their last infusion of an allogenic CAR T cell product.

ELIGIBILITY:
Inclusion Criteria:

* Received an allogenic CAR T-cell product infusion to treat an oncologic condition in a previous Allogene or Servier sponsored clinical study

Exclusion Criteria:

* Less than 12 months of follow up after the last allogeneic CAR T-cell product, unless approved by the Allogene Medical Monitor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have received an allogeneic CAR T-cell product.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2039-01 (Estimated); Study Completion 2039-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed adverse events potentially related to allogeneic CAR T-cell product and allogeneic CAR T-cell product-related SAEs | Up to 15 years post treatment with allogeneic CAR T-cell product
Overall survival (OS) | Up to 15 years post treatment with allogeneic CAR T cell product
Presence of replication competent lentivirus (RCL) in blood | Up to 15 years post treatment with allogeneic CAR T cell product

CONTACTS AND LOCATIONS:
Overall Officials: Allogene Study Director, Study Director — Allogene Therapeutics, Inc.
Locations (1):
- Circuit Clinical, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No